CLINICAL TRIAL: NCT00523939
Title: Phase II Study of Intrathecal Therapy With DepoCyt for Active Lymphomatous or Leukemic Meningitis
Brief Title: DepoCyt for Active Lymphomatous or Leukemic Meningitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: Duke University (Other)
Collaborators: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00009742
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Results first posted 2011-03-14 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2012-11

CONDITIONS: Neoplastic Meningitis; Lymphoma, B Cell
Keywords: Lymphoma; Leukemia; Leukemic Meningitis; Lymphomatous Meningitis
MeSH Terms: conditions — Meningeal Carcinomatosis; Lymphoma, B-Cell; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lymphomatous (Experimental): Subjects with Lymphomatous Meningitis
  Interventions: Drug: cytarabine liposome injection
- Leukemic (Experimental): Subjects with Leukemic Meningitis
  Interventions: Drug: cytarabine liposome injection

INTERVENTIONS:
Drug: cytarabine liposome injection — 50 mg intrathecal every 14 days for 8 doses, then every 28 days for six doses
  Other Names: DepoCyt

SUMMARY:
The purpose of this study is to determine the response rate of lymphomatous meningitis or leukemic meningitis to DepoCyt. The safety of DepoCyt, the number of people who respond well to the study drug, and the response of symptoms to the study drug will also be determined.

DETAILED DESCRIPTION:
DepoCyt is a sustained-release formulation of the chemotherapy drug, cytarabine (Ara-C), which is used for the treatment of patients with lymphomatous or leukemic meningitis, a complication of lymphoma/leukemia that is characterized by the spread of cancer to the central nervous system.

DepoCyt is introduced into the spinal fluid, through a needle inserted into the spinal canal or through a reservoir placed under the scalp by a neurosurgeon. DepoCyt will be given every two weeks i.e. week 1 and week 3 initially. After the second dose, a lumbar puncture will be done to check the spinal fluid for cancer cells. If there has been a good response, DepoCyt will be given every 14 days for 6 doses i.e., weeks 5, 7, 9, 11, 13, 15 and then every 28 days for six doses i.e., weeks 19, 23, 27, 31, 35, and 39. Blood tests and lumbar punctures will be done throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically confirmed, or radiographic evidence for lymphomatous or leukemic meningitis. If the CSF cytology is negative, patients must have MRI/CT brain and clinical findings consistent with neoplastic meningitis.
* Karnofsky Performance Score of 60 or above.
* Age ≥ 18 years.
* Patients must have adequate hematologic, renal and liver function. Laboratory
* Absolute neutrophil count (ANC) ≥ 1,500/mm3 or white blood cell count > 3,000/mm3
* Platelet count ≥ 100, 000/mm3
* BUN and serum creatinine must be ≤ 1.5 times upper limit of laboratory normal
* Total and direct serum bilirubin must be ≤ 1.5 times upper limit of laboratory normal
* SGOT and SGPT ≤ 3.0 times upper limit of laboratory normal
* Alkaline phosphatase derived from liver ≤ 2.0 times upper limit of laboratory normal
* No uncontrolled infection other than human immunodeficiency virus that is being treated with anti-retroviral therapy
* Patients who have had prior CNS radiation, prior intrathecal methotrexate, and prior CNS prophylaxis with intrathecal or intravenous cytarabine or methotrexate are eligible
* Written informed consent

Exclusion Criteria:

* Experimental/Investigational chemotherapy, immunotherapy, or biologic therapy within four weeks prior to study
* Concurrent systemic chemotherapy with high dose methotrexate, high dose cytarabine, or high dose thiotepa (they cross the blood brain barrier at high levels)
* Patients receiving whole brain radiotherapy or craniospinal irradiation
* Previous (less than 2 years from diagnosis) or concurrent malignancies at other sites with the exception of fully treated carcinoma in situ of the cervix, basal cell carcinoma of the skin, and squamous cell carcinoma of the skin, or prostate cancer not requiring ongoing chemotherapy
* Pregnant or lactating women
* Known active meningeal infection
* Evidence of obstructive hydrocephalus requiring neurosurgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Rizzieri, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment June 2006 - September 2008. Study stopped early due to poor accrual.
Period: Overall Study
Arm/Group | Lymphomatous | Leukemic
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lymphomatous | Leukemic | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To evaluate response rate using intrathecal DepoCytTM in two cohorts of patients, one with active lymphomatous meningitis and another with active leukemic meningitis.
Time Frame: 1 year
Population: Primary outcome measure was not assessed due to early study termination.
Arm/Group | Lymphomatous | Leukemic
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Time to Neurologic Progression
Time Frame: 2 years
Arm/Group | Lymphomatous | Leukemic
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- All Subjects: Subjects with Lymphomatous or Leukemic Meningitis.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 3/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=4)
Death not associated with CTCAE term, disease progression (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Arachnoiditis (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=4)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Slurred speech (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (2) — Thrombocytopenia
Rash (Skin and subcutaneous tissue disorders) | 1 (1) — Folliculitis
Seizure (Nervous system disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) — Possible seizure
DVT (Vascular disorders) | 1 (1)
Mood alteration (Nervous system disorders) | 2 (2)
Pain (General disorders) | 1 (3)
Edema (General disorders) | 1 (1)
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

LIMITATIONS AND CAVEATS:
Adverse events for both arms, lymphomatous and leukemic, were combined due to low accrual and early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes